CLINICAL TRIAL: NCT03168659
Title: Post-Approval Study of the HeartLight Endoscopic Ablation System for the Treatment of Atrial Fibrillation
Brief Title: CardioFocus HeartLight Post-Approval Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CardioFocus (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-3944
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (Other): Pulmonary vein isolation ablation with HeartLight Endoscopic Ablation System
  Interventions: Device: HeartLight; Procedure: Ablation

INTERVENTIONS:
Device: HeartLight — HeartLight Endoscopic Ablation System
Procedure: Ablation — Pulmonary vein isolation ablation

SUMMARY:
This is a post-approval study to evaluate the clinical outcomes in a cohort of participants treated during commercial use of the HeartLight System to confirm results of the previously conducted pivotal clinical study.

DETAILED DESCRIPTION:
This is a prospective, open-label, multi-center, single arm study designed to assess continued safety and effectiveness of the HeartLight System during commercial use in participants being treated for drug refractory, symptomatic, paroxysmal atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* planned for catheter ablation due to symptomatic paroxysmal atrial fibrillation
* failure of at least one anti-arrhythmic drug
* others

Exclusion Criteria:

* overall good health as established by multiple criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2017-06-16 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants free from symptomatic atrial fibrillation (AF) or symptomatic atypical atrial flutter/atrial tachycardia (AFL/AT) lasting longer than 30 seconds post the 90 day blanking period | Day 91 through 12 months
  The outcome will be assessed from 91 days post procedure through 12 months

OTHER OUTCOMES:
Chronic Effectiveness | 36 months
  Freedom from symptomatic AF or symptomatic atypical AFL/AT
Chronic Safety | 36 months
  Reporting of adverse events
Effect of Operator Experience on primary effectiveness endpoint | 36 months
  Assess relationship between operator experience and freedom from symptomatic AF or symptomatic atypical AFL/AT
Effect of Operator Experience on primary safety endpoint | 36 months
  Assess relationship between operator experience and rate of Primary Adverse Events (PAE)
Safety Outcomes by Gender | 12 months and 36 months
  Assess relationship between gender and rate of PAEs
Neurological Events | 36 months
  Assess relationship between neurological events and procedural parameters

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Arizona Sarver HeartCenter, Tucson, Arizona
  - University of Illinois, Chicago, Illinois
  - Mount Sinai Hospital, New York, New York
  - University Of Virginia Health System, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No